CLINICAL TRIAL: NCT02399540
Title: Late LTP-like Plasticity Effects of tDCS in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Rick van der Vliet, MSc, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEC-2014-203
Record Dates: First submitted 2015-03-15; First posted 2015-03-26 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Stroke; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sham (Sham Comparator): Day 1: sham stimulation Day 2: sham stimulation
  Interventions: Device: Sham
- Conventional Paired tDCS (Active Comparator): Day 1: sham stimulation Day 2: conventional tDCS
  Interventions: Device: Conventional Paired tDCS
- Conventional Unpaired tDCS (Active Comparator): Day 1: conventional tDCS Day 2: sham stimulation
  Interventions: Device: Conventional Unpaired tDCS
- Late LTP-like Plasticity tDCS (Experimental): Day 1: late LTP-like Plasticity tDCS Day 2: sham stimulation
  Interventions: Device: Late LTP-like Plasticity tDCS

INTERVENTIONS:
Device: Sham — Bihemispheric 1mA Sham protocol: sham - pause - sham
  Arms: Sham
Device: Conventional Paired tDCS — Bihemispheric 1mA Sham protocol: sham - pause - sham Conventional Paired tDCS protocol: 20 minutes tDCS - pause - sham
  Arms: Conventional Paired tDCS
Device: Conventional Unpaired tDCS — Bihemispheric 1mA Sham protocol: sham - pause - sham Conventional Unpaired tDCS protocol: 20 minutes tDCS - pause - sham
  Arms: Conventional Unpaired tDCS
Device: Late LTP-like Plasticity tDCS — Bihemispheric 1mA Sham protocol: sham - pause - sham Late LTP-like Plasticity tDCS protocol: 10 minutes tDCS - 25 minutes pause - 10 minutes tDCS
  Arms: Late LTP-like Plasticity tDCS

SUMMARY:
Rationale: About 80% of stroke patients suffer motor impairments, but current therapies have limited effects on motor recovery. Therefore, investigating new potential therapeutic approaches is crucial. Transcranial Direct Current Stimulation (tDCS) is a form of non-invasive electrical stimulation where a weak current is applied through electrodes over the scalp. This stimulation is known to (1) induce changes in neuronal excitability -which can last up to one day with late LTP-like plasticity protocols- in a polarity and site-specific manner, and (2) facilitate motor learning and stroke recovery. However, it is unknown how the motor cortex excitability changes that follow tDCS relate to the increase in motor learning and recovery potential. The currently upheld hypothesis is that motor learning needs to be synchronized in time with electrical stimulation (paired stimulation), but recent results from our lab suggest that tDCS also increases skill learning after stimulation has ended (unpaired stimulation). If this is true, tDCS has a much larger therapeutic window and is a more valuable clinical tool than currently believed. Therefore, the investigators want to investigate how late LTP-like plasticity tDCS affects the increase in skill learning normally seen with tDCS when applied 24 hours before training. The outcome of this study can provide important guidelines on effective motor therapy during stroke rehabilitation.

Objective: Identify the effect of late LTP-like plasticity tDCS in chronic stroke patients on skill learning 24 hours later.

Study design: Double-blinded, randomized between-subjects trials. Study population: Chronic stroke patients. Main study parameters/endpoints: The main objective of the study is to determine the effect of late LTP-like plasticity tDCS on skill learning 24 hours later. As a motor learning paradigm, the investigators will use a circuit tracking task which chronic stroke patients perform better if tDCS is applied concurrently. During this task, patients have to trace a cursor over a circuit as fast and accurately as possible by moving a computer mouse. Skill will be quantified by calculating a combined speed/ accuracy score and skill improvement compared to baseline (LI; the learning index) will be compared between the sham, conventional unpaired tDCS, conventional paired tDCS groups and the late LTP-like plasticity tDCS groups.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (> 6 months) stroke patient
* Aged 18-79 years
* Motor deficit in the upper limb due to the stroke

Exclusion Criteria:

* Absence of recordable MEPs from the ADM after TMS
* Absence of voluntary movement (Fugl-Meyer < III)
* Head injury or the presence of intracranial metal or intracranial lesions
* History of cranial irradiation
* History of epilepsy
* Presence of a pacemaker
* Taking anticonvulsant or neuroleptic medication
* Substance abuse
* Inability to understand instructions
* History of psychiatric disorders

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Motor Skill Retention | Day 9
  Motor skill retention will be assessed on the circuit game

SECONDARY OUTCOMES:
Maximum Grip Force | Day 1 and Day 9
  Maximum Grip Force will be assessed using a Jamar Dynamometer
Purdue Pegboard Test | Day 1 and Day 9

CONTACTS AND LOCATIONS:
Locations (1):
- Rijndam, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Result] Lefebvre S, Laloux P, Peeters A, Desfontaines P, Jamart J, Vandermeeren Y. Dual-tDCS Enhances Online Motor Skill Learning and Long-Term Retention in Chronic Stroke Patients. Front Hum Neurosci. 2013 Jan 9;6:343. doi: 10.3389/fnhum.2012.00343. eCollection 2012. PMID 23316151
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- [Derived] van der Vliet R, Ribbers GM, Vandermeeren Y, Frens MA, Selles RW. BDNF Val66Met but not transcranial direct current stimulation affects motor learning after stroke. Brain Stimul. 2017 Sep-Oct;10(5):882-892. doi: 10.1016/j.brs.2017.07.004. Epub 2017 Jul 13. PMID 28751226